CLINICAL TRIAL: NCT01506804
Title: The Efficacy of Exercise Therapy Followed by Ultrasound Guided Injection in Patients With a Painful Shoulder - a Randomised Controlled Study With Blinded Observer
Brief Title: Exercise Therapy and Ultrasound Guided Injections in Painful Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Collaborators: Oak Foundation (Other); The Danish Physiotherapy Foundation (Unknown); Fund for Physiotherapy in Private Practice (Unknown); Aase and Ejnar Danielsens Foundation (Other)
Responsible Party: Principal Investigator, Henning Bliddal, Professor, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-4-2010-002
Record Dates: First submitted 2011-05-05; First posted 2012-01-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Shoulder Bursitis
Keywords: Shoulder; Impingement; Ultrasound; injection of glucocorticosteroid; exercise
MeSH Terms: conditions — Motor Activity | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training of painful shoulder (Experimental): Steroid injection X 2 and 10 weeks exercise program of painful shoulder
  Interventions: Other: methylprednisolone
- Contralateral training (Placebo Comparator): Steroid injection X 2 and 10 weeks exercise program of asymptomatic shoulder
  Interventions: Other: methylprednisolone

INTERVENTIONS:
Other: methylprednisolone — Steroid injection X 2 and 10 weeks exercise program of painful shoulder vs exercise program of contralateral shoulder

SUMMARY:
Many patients experience an effect of steroid injection, however the effect is often short lasting and recurrence of symptoms is common. The short term effect of injection has been shown to be much better than exercise therapy; however over time the superior effect of injection compared to exercise does not last. Injection in combination with exercise therapy might be a more sufficient therapy than injection alone. The aim of this study is to investigate a combination of steroid injection and a 10 week exercise program. In addition, the study tests the validity of clinical impingement tests using ultrasound verified impingement as gold standard.

DETAILED DESCRIPTION:
For many patients unspecific pain and reduced motion in the shoulder is a common complaint. It is believed that the main reason for shoulder pain comes from inflammation of the bursa.

Many patients experience an effect of steroid injection, however the effect is often short lasting and recurrence of symptoms is common. Exercise therapy for the muscles around the shoulder joint is also common treatment for shoulder pain. The short term effect of injection has been shown to be much better than exercise therapy; however over time the superior effect of injection compared to exercise does not last. The anti-inflammatory and pain releasing effect of steroid injection in combination with exercise therapy increasing the strength and control of the muscles around the shoulder joint, might be a more sufficient therapy than injection alone. Thus, the aim of this study is to investigate a combination of steroid injection and a 10 week exercise program in patients with a painful shoulder.

Many different clinical tests are used to examine the pathological compression of the bursa during motion in the shoulder joint (impingement). However, it is actually not known if the pain in motion is caused by compression of the bursa. Part of this study therefore is to test the validity of clinical impingement tests using ultrasound verified impingement as gold standard.

Studies comparing injection given guided by ultrasound to blind injections have shown that the ultrasound guided injections are more likely to place the active stuff correctly in the swollen bursa. In this study all injections will be given ultrasound guided. In the ultrasound examination the thickness of the bursa will be measured in all patients in order to investigate if swollenness of the bursa can explained the pain and dysfunction of the shoulder joint

ELIGIBILITY:
Inclusion Criteria:

* Pain and reduced motion in the shoulder for more than four weeks
* Ultrasound verified swollenness of the bursa.

Exclusion Criteria:

* Bilateral pain in the shoulder joints
* Rupture of the rotator cuff or biceps tendons
* Generalised disease which can explain the shoulder pain
* OA in the shoulder joint
* Diabetes
* Positive compression test of the cervical spine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-11; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pain in the shoulder in both rest and motion (VAS) | 6 months

SECONDARY OUTCOMES:
Ultrasound | 6 months
Strength | 6 months
Clinical impingement | 6 months
Shoulder function | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bliddal, Professor, Principal Investigator — The Parker Institute, University of Copenhagen
Locations (1):
- The Parker Institute, Frederiksberg Hospital, Frederiksberg, Denmark

REFERENCES:
- [Derived] Ellegaard K, Christensen R, Rosager S, Bartholdy C, Torp-Pedersen S, Bandholm T, Danneskiold-Samsoe B, Bliddal H, Henriksen M. Exercise therapy after ultrasound-guided corticosteroid injections in patients with subacromial pain syndrome: a randomized controlled trial. Arthritis Res Ther. 2016 Jun 4;18(1):129. doi: 10.1186/s13075-016-1002-5. PMID 27262892
- See also: The Parker Institute, Copenhagen — http://www.parkerinst.dk